CLINICAL TRIAL: NCT07012655
Title: Color Doppler Ultrasonography Evaluation of Abdominal and Peripheral Vasculopathy in Systemic Sclerosis Patients
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Farrag Ahmed Mohamed, Lecturer of Rheumatology and Rehabilitation, Assiut University
Other Study IDs: SFA12025
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; Doppler Ultrasound
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Colour Doppler Ultrasound — All study participants will undergo abdominal Ultrasound and Colour doppler ultrasound study of the superior and inferior mesenteric arteries and the resistance index and peak systolic velocity (cm/s) of radial and ulnar arteries measured by ultrasonography color Doppler with spectral wave analysis.

SUMMARY:
In the current study we aim to assess the macrovascular involvement in SSc patients through an ultrasound (US) evaluation of radial and ulnar arteries and splanchnic vessels.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a connective tissue disease (CTD) characterized by diffuse cutaneous sclerosis of skin and organs, small vessel vasculopathy and immune system dysregulation associated with the production of autoantibodies.

Although small vessel vasculopathy can be considered a hallmark of this disease, large vessels can also be involved. Accordingly, involvement of medium vessels such as the ulnar artery has been evaluated in the literature, with results showing how ulnar artery occlusion (UAO) could be considered as a severity marker of vasculopathy as well as a predictive marker of digital ulcers (DUs), which are typically more frequent in patients with limited cutaneous (lc) SSc.

The gastrointestinal (GI) tract is one of the most frequently involved organs, affecting the majority (75-90%) of SSc patients.

GI involvement is often largely asymptomatic because it is frequently subclinical until severe tissue damage occurs. Once symptoms occur, SSc-related GI involvement heavily impacts morbidity and mortality, with patients experiencing significant emotional and social burdens and decreased survival in severe cases.

Unfortunately, the diagnosis of GI involvement is challenging because it is often delayed by the paucity of signs and symptoms early in the disease. Moreover, several diagnostic investigations that are useful in defning GI involvement are either invasive, expensive or not very informative.

Understanding the etiology and early phases of GI involvement, therefore, remains a high priority in SSc research. The aim would be to identify patients at high risk of developing progressive GI involvement, monitor disease activity, in the vessels or other relevant tissues, and intervene before the development of signifcant damage/dysfunction.

Bandini et al. showed how potentially the splanchnic vessels in SSc may be non-invasively investigated with abdominal US and color Doppler US, showing that some morphological and functional US parameters of mesenteric arteries of SSc patients are different from healthy controls defining a "bowel vasculopathy".

Abdominal ultrasound (US) is a unique tool that allows for the noninvasive assessment of the vasculature and major parts of the GI tract, including extra-intestinal features and splanchnic vessels as well as peripheral vessels.

ELIGIBILITY:
Inclusion Criteria:

* Adult systemic sclerosis patients fulfilling the criteria for the diagnosis by American College of Rheumatology /European league against rheumatism 2013 classification criteria for systemic sclerosis, who accept to participate in the current study.

Exclusion Criteria:

* Individuals with other autoimmune diseases (rheumatoid arthritis, dermatomyositis, mixed connective tissue disease).
* those who Refuse to participate in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 50 participants:
  Group 1: 25 Adult Systemic sclerosis fulfilling the criteria for the diagnosis by American College of Rheumatology /European league against rheumatism 2013 classification criteria for systemic sclerosis.
  Group 2: 25 healthy matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Macro vascular involvement in systemic sclerosis patients | day 1
  Assess the macro vascular involvement in SSc patients through an ultrasound (US) evaluation of radial and ulnar arteries and splanchnic vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Farrag, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lescoat A, Coiffier G, Rouil A, Droitcourt C, Cazalets C, de Carlan M, Perdriger A, Jego P. Vascular Evaluation of the Hand by Power Doppler Ultrasonography and New Predictive Markers of Ischemic Digital Ulcers in Systemic Sclerosis: Results of a Prospective Pilot Study. Arthritis Care Res (Hoboken). 2017 Apr;69(4):543-551. doi: 10.1002/acr.22965. Epub 2017 Mar 3. PMID 27390194
- [Background] Romano E, Rosa I, Fioretto BS, Matucci-Cerinic M, Manetti M. Increased Circulating Soluble Junctional Adhesion Molecules in Systemic Sclerosis: Association with Peripheral Microvascular Impairment. Life (Basel). 2022 Nov 4;12(11):1790. doi: 10.3390/life12111790. PMID 36362943